CLINICAL TRIAL: NCT00256360
Title: A Randomized Phase II Trial Exploring Feasibility of Densification and Optimal Sequencing of Postoperative Adjuvant Fluorouracil, Epirubicin Plus Cyclophosphamide (FEC) and Docetaxel Chemotherapy in Patients With High Risk Primary Operable Breast Cancer
Brief Title: Trial Exploring Feasibility of Densification and Optimal Sequencing of Postoperative Adjuvant Fluorouracil, Epirubicin Plus Cyclophosphamide (FEC) and Docetaxel Chemotherapy in Patients With High Risk Primary Operable Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: St-Augustinus Wilrijk (Unknown)
Responsible Party: Principal Investigator, prof. dr. Hans Wildiers, adjunct head of clinic, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-001876-11
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; adjuvant; dose dense; docetaxel; pegfilgrastim
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim

INTERVENTIONS:
Drug: dose dense with neulasta

SUMMARY:
The rationale of this randomized phase II study is to investigate the feasibility of sequenced densified FEC and docetaxel based regimens in patients with primary operable high-risk breast cancer. Several phase III and phase II clinical trials showed the benefits of dose-dense therapy (Q2W) over conventional treatment in breast cancer, lymphoma and SCLC. The aim of the study is also to demonstrate that further shortening of treatment interval from 14 days to 10-11 days in FEC regimen is feasible and will not compromise patient's safety. The results of this randomized phase II study should serve as a basis for follow-up randomized phase III trial comparing conventional versus densified sequential FEC and docetaxel based regimens.

DETAILED DESCRIPTION:
Arm A:

The three cycles of conventional FEC followed by three cycles of docetaxel regimen will be given at the following doses:

Fluorouracil 500 mg/m² by i.v. bolus or infusion, Epirubicin 100 mg/m² by 30 minutes i.v. infusion and Cyclophosphamide 500 mg/m² by i.v. bolus or infusion followed by docetaxel 100 mg/m2 i.v. infusion. All drugs will be administered intravenously on Day 1 of each 21-day cycle without support of growth factors.

Pegfilgrastim is only allowed in secondary prophylaxis: febrile neutropenia or prolonged grade IV neutropenia. In the event of febrile neutropenia or prolonged grade IV neutropenia, pegfilgrastim or filgrastim is given for treatment, and pegfilgrastim should be further administered on day 2 of each subsequent cycle of chemotherapy.

The total duration of treatment is 18 weeks.

Arm B:

The three cycles of conventional docetaxel followed by three cycles of FEC regimen will be given at the following doses:

Docetaxel 100 mg/m2 i.v. infusion followed by Fluorouracil 500 mg/m² by i.v. bolus or infusion, Epirubicin 100 mg/m² by 30 minutes i.v. infusion and Cyclophosphamide 500 mg/m² by i.v. bolus or infusion. All drugs will be administered intravenously on Day 1 of each 21-day cycle without support of growth factors.

Pegfilgrastim is only allowed in secondary prophylaxis: febrile neutropenia or prolonged grade IV neutropenia. In the event of febrile neutropenia or prolonged grade IV neutropenia, pegfilgrastim or filgrastim is given for treatment, and pegfilgrastim should be further administered on day 2 of each subsequent cycle of chemotherapy.

The total duration of treatment is 18 weeks.

Arm C:

The four cycles of dose-dense FEC followed by four cycles dose-dense docetaxel regimen will be given at the following doses:

Fluorouracil 375 mg/m² by i.v. bolus or infusion, Epirubicin 75 mg/m² by 30 minutes i.v. infusion and Cyclophosphamide 375 mg/m² by i.v. bolus or infusion followed by docetaxel 75 mg/m2. FEC regimen will be administered intravenously on Day 1 of each 10-11-day cycle and docetaxel will be given on Day 1 of each 14-day cycle.

Pegfilgrastim (Neulasta) fixed dose of 6 mg (0.6 mL of a 10 mg/mL solution) as a single subcutaneous injection will be given in on Day 2 of each study cycle.

The total duration of treatment is 14 weeks.

Arm D:

The four cycles of dose-dense docetaxel followed by four cycles dose-dense FEC regimen will be given at the following doses:

Docetaxel 75 mg/m² followed Fluorouracil 375 mg/m² by i.v. bolus or infusion, Epirubicin 75 mg/m² by 30 minutes i.v. infusion and Cyclophosphamide 375 mg/m² by i.v. bolus or infusion. Docetaxel will be given on Day 1 of each 14-day cycle and FEC regimen will be administered intravenously on Day 1 of each 10-11-day cycle.

Pegfilgrastim (Neulasta) fixed dose of 6 mg (0.6 mL of a 10 mg/mL solution) as a single subcutaneous injection will be given on Day 2 of each study cycle.

The total duration of treatment is 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven early breast cancer requiring adjuvant chemotherapy (lymph node positive or other features of high risk according to St-Gallen criteria)
* Margins of resection histologically free of invasive carcinoma and ductal carcinoma in situ.
* Radiotherapy performed according to center's policy and always follows completion of adjuvant chemotherapy
* Performance status 0 to 1 on the ECOG scale (Appendix A)
* The determination of ER and PgR is mandatory (immunohistochemical methods required; ER and/or PgR positivity is defined as > 1% of positive cells). Also determination of Her2neu is mandatory, either by immunohistochemistry or by FISH
* Age > 18 years and age <70 years (upper age limit based on the lack of safety data for this population).
* Normal cardiac function (assessment of LVEF by MUGA scan or echocardiography above the lower limit of normal for the institution).
* Adequate organ function (as defined by neutrophils > 1.5 x109/L, Platelets > 100 x 109/L, Hemoglobin > 10 g/dl, total bilirubin > 1 UNL, ASAT (SGOT) and ALAT (SGPT) > 1.5 UNL, alkaline phosphatase > 2.5 UNL, creatinine > 1.5 mg/dl (150 µmol/L)
* Complete staging work-up within 2 months prior to registration. All patients will have bilateral mammography, chest X-ray (PA and lateral) and/or CT-scan, abdominal ultrasound and/or CT scan, bone scan. In case of positive bone scan suspicious for metastases, bone X-ray (or bone CT-scan on spinal hot spots) is mandatory to rule out the possibility of metastatic disease. Other tests may be performed as clinically indicated.
* Negative pregnancy test (urine or serum) within 7 days prior to registration for all women of childbearing potential. Patients of childbearing potential must implement adequate non-hormonal measures to avoid pregnancy during study treatment (chemotherapy, radiotherapy and endocrine therapy). No pregnant or lactating patients are allowed.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion criteria:

* Metastatic disease (M1) or inoperable residual axillary disease
* Prior systemic anticancer therapy for breast cancer (chemotherapy, hormone therapy of immunotherapy)
* Prior radiation therapy for breast cancer.
* Pre-existing motor or sensory neurotoxicity of a severity > grade 2 by NCI criteria.
* Pregnant or lactating patients
* Other serious illness or medical condition:
* Congestive heart failure or unstable angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or high-risk uncontrolled arrhythmias.
* History of significant neurological or psychiatric disorders that would prohibit the understanding and giving of informed consent.
* Active uncontrolled infection
* Active peptic ulcer, unstable diabetes mellitus.
* Past or current history of other neoplasm except for curatively treated basal cell skin cancer or in situ carcinoma of the cervix.
* Chronic treatment with steroids unless initiated > 6 months prior to study entry and at low dose (< 20 mg methylprednisolone or equivalent)
* Concurrent treatment with hormonal replacement therapy: this treatment should be stopped at least 15 days before study entry.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117
Dates: Start 2005-09; Study Completion 2006-05

PRIMARY OUTCOMES:
To assess the feasibility of FEC and docetaxel based sequential regimens given in dose-dense fashion (FEC every 10-11 days and docetaxel every 14 days) with pegfilgrastim in patients with high-risk primary breast cancer.

SECONDARY OUTCOMES:
To assess the safety and tolerability of FEC and docetaxel regimens including (febrile) neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: Hans Wildiers, MD, PhD, Principal Investigator — UZ Gasthuisberg Leuven
Locations (1):
- UZ Gasthuisberg Leuven, Leuven, Belgium